CLINICAL TRIAL: NCT05661474
Title: The Effects of Fitostimoline® Hydrogel Versus Saline Gauze Dressing in Patients With Diabetic Foot Ulcers: a Monocentric, Two-arm, Open-label, Randomized, Controlled Trial.
Brief Title: Fitostimoline® Hydrogel Versus Saline Gauze Dressing in Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Prof, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 350/20
Record Dates: First submitted 2022-12-12; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; dressing; medication
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fitostimoline® hydrogel group (Experimental): Participant randomized to the Fitostimoline® hydrogel group underwent sharp surgical debridement at each visit (every 2 weeks) to remove necrotic tissue and slough. After debridement operation, was performed disinfection with povidone-iodine, and cleansing with sterile saline solution. Then was applaied Fitostimoline ® hydrogel, finally the wound was covered with gauze.
  Interventions: Drug: Fitostimoline ® hydrogel group
- Saline gauze group (Active Comparator): Participant randomized to the Saline gauze group underwent sharp surgical debridement at each visit (every 2 weeks) to remove necrotic tissue and slough. After debridement operation, was performed disinfection with povidone-iodine, and cleansing with sterile saline solution. Then was applaied saline gauze, finally the wound was covered with gauze.
  Interventions: Drug: Saline gauze group

INTERVENTIONS:
Drug: Fitostimoline ® hydrogel group — Treatment of DFUs with Fitostimoline® hydrogel every day for 12 weeks.
  Arms: Fitostimoline® hydrogel group
Drug: Saline gauze group — Treatment of DFUs with saline gauze every day for 12 weeks.
  Arms: Saline gauze group

SUMMARY:
Diabetes Mellitus (DM) is one of the most widespread metabolic diseases and the alarming rise in its prevalence worldwide poses enormous challenges. The microvascular and macrovascular complications of DM heavy impact on longevity and quality of life, and in particular diabetic foot ulcers (DFUs) are among the ten top causes of worldwide disease burden and disability Essential components of the standard care, management, and treatment of DFUs are represented by health education, strict control of blood glucose and cardiovascular risk factors, offloading, local debridement, and adequate dressing. A wide variety of dressing is available, and these include basic contact dressings (low adherence dressings such as saline gauze, paraffin gauze or simple absorbent dressings) and advanced dressings (alginate, hydrogel, films, hydrocolloid, foam).

It is important underline that due to lack of evidence from head-to-head randomized controlled trials (RCTs), the relative effects of any of these dressings in DFUs remain unclear. Consequently, so far clinical evidence supporting the choice for either hydrogel or saline gauze dressing, has been related mostly on clinician perception rather than high quality evidence. Here we evaluated the efficacy and safety of Fitostimoline® hydrogel dressing versus saline gauze dressing in patients with DFUs in a monocentric, two-arm, open-label, randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes and type 2 diabetes,
* adult patients with DFUs at Grades IC or IIC for a period of at least 12 weeks,
* an akle brachial index >0.8,
* be able to understand simple instructions,
* provided voluntary, signed informed consent

Exclusion Criteria:

* active infection
* evidence of ischaemia in the limb,
* osteomyelitis,
* gangrene,
* systemic inflammatory or autoimmune disease,
* use of corticosteroids, immunosuppressive agents, radiation therapy and chemotherapyan,
* known hypersensitivity to any of the dressing components.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients complete responders | 12 weeks
  The primary outcome was the proportion of patients that at the end of study period of 12 weeks (V6) were categorized as complete responders -complete healing of the wound defined as reepithelialisation of 100% without medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Medicine and Surgery Federico II University, Naples, Italy